CLINICAL TRIAL: NCT01051284
Title: A Pilot Study of Full Dose Gemcitabine and Hypofractionated Stereotactic Radiosurgery in the Treatment of Unresectable Pancreatic Cancer
Brief Title: A Study of Gemcitabine and Cyberknife Radiation Therapy for Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Michael J Pishvaian, Assistant Professor, Georgetown University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-169
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; Newly diagnosed; Cyberknife; Gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyberknofe and Gemcitabine (Experimental): Cyberknife radiation and 6 cycles Gemcitabine
  Interventions: Radiation: Cyberknife radiation and gemcitabine

INTERVENTIONS:
Radiation: Cyberknife radiation and gemcitabine — 25 Gray of radiation will be given in 5 fractions using the Cyberknife Gemcitabine 1000 mg/m2 intravenously will be given once a week on days 1, 8, and 15 of every 28-day cycle for 6 cycles
  Other Names: Gemcitabine; Gemzar

SUMMARY:
People with pancreatic cancer that cannot be cured by surgery are being asked to participate in this study.

The purpose of this study is to test the ability of the radiation oncologists to administer Cyberknife therapy along with Gemcitabine chemotherapy for patients with pancreatic cancer. Radiation and Gemcitabine are both effective at killing cancer cells but they generally cannot be given at the same time. Cyberknife therapy is highly focused radiation that is being used extensively at Georgetown University and around the United States to treat a number of cancers. It is believed that because Cyberknife is so highly focused it can be given safely with regular doses of chemotherapy to attack cancer cells in two ways at the same time.

This research is being done because it is not known if using Cyberknife with chemotherapy will be a safe way to treat pancreatic cancer.

DETAILED DESCRIPTION:
This is a single arm, open-label pilot study of Cyberknife plus Gemcitabine in 10 patients with locally advanced pancreatic cancer who have not received prior local or systemic therapy for their pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven unresectable, non-metastatic pancreatic adenocarcinoma with measurable or evaluable disease and without involvement of the duodenum
* Performance Status 0-2
* No prior anticancer therapy for pancreatic adenocarcinoma
* No prior anticancer therapy of any kind within the last 5 years
* Adequate hepatic, bone marrow, and renal function
* Life expectance of > 12 weeks
* Women of childbearing potential must have a negative serum pregnancy test

Exclusion Criteria:

* Duodenal involvement of pancreatic cancer
* Metastatic cancer
* Active severe infection, or known chronic infection with HIV, hepatitis B virus, or hepatitis C virus
* Cardiovascular disease including unstable angina, therapy for life-threatening ventricular arrhythmia, myocardial infarction, stroke, or congestive heart failure within the last 6 months
* Life-threatening visceral disease or other severe concurrent disease
* Pregnant or breastfeeding
* Anticipated patient survival under 3 months
* Another active malignancy within the past 5 years except for cervical cancer in situ, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To demonstrate that radiation treatments can be reproduced as determined by evaluation of the prescription isodose curves | 10 days

SECONDARY OUTCOMES:
Acute and late toxicity as determined by patient self-reporting instruments that assess gastrointestinal side effects | 6 months
Quality of life as determined by patient self-reporting instruments | 6 months
Acute stomach/duodenal mucosa injury as assessed by upper endoscopy | one month
Late stomach/duodenal mucosa injury as assessed by upper endoscopy | 6 months
Feasibility of integrating metabolomic analysis into the evaluation of patients with unresectable pancreatic cancer undergoing chemotherapy and radiation therapy measured by the ability to collect tumor specimens | 6 months
The feasibility of measuring pancreatic cancer stem cell populations by analysis of fine needle aspirate specimens | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Pishvaian, MD, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States